CLINICAL TRIAL: NCT06637852
Title: Sexual and Urinary Function Improvement for Cancer Survivors- Promoting Access to Collaborative Treatment (SUFICS-PACT)
Brief Title: Sexual and Urinary Function Improvement for Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-00945
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Urinary Dysfunction; Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUFICS-PACT (Experimental): The Sexual and Urinary Function Improvement for Cancer Survivors- Promoting Access to Collaborative Treatment (SUFICS-PACT) intervention integrates a collaborative care model in primary care to facilitate problem identification, comprehensive treatment, and close follow-up for sexual and urinary dysfunction.
  Interventions: Behavioral: SUFICS-PACT
- Usual care (No Intervention): Participants assigned to this group will continue with usual care.

INTERVENTIONS:
Behavioral: SUFICS-PACT — SUFICS-PACT includes sexual and urinary dysfunction screening, collaborative treatment of sexual and urinary dysfunction, and care managers who are mental health professionals with training in psychosexual counseling. Mental health professionals will facilitate a comprehensive approach to sexual dysfunction, as emphasized by the biopsychosocial model of sexual health. SUFICS-PACT also emphasizes close follow up, which is important for sexual function recovery after prostate cancer treatment.
  Arms: SUFICS-PACT

SUMMARY:
The purpose of this study is to test the efficacy of SUFICS-PACT to identify and treat sexual and urinary dysfunction in prostate cancer survivors at NYC H+ H/Bellevue, the oldest public hospital in the US. This study will evaluate the implementation of an adapted sexual and urinary function collaborative care model at NYC Health+Hospitals/Bellevue. The study will test the efficacy of this collaborative care model through a randomized controlled trial in the adult primary care clinic; the intervention arm will receive collaborative treatment consisting of a care manager who has specialty training in mental health and psychosexual counseling, a primary care nurse practitioner who leads symptom management, primary care physicians who supervise the team, and a team specialty consult liaison.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Have a diagnosis of prostate cancer
* Have sought care/treatment for prostate cancer

Exclusion Criteria:

* Patients under 18 years old
* Patients who have not sought care/treatment for prostate cancer
* Patients who are categorized as "vulnerable subjects," such as minors or incarcerated individuals.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients identified and treated for sexual dysfunction | Year 5
Number of patients identified and treated for urinary dysfunction | Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Nnenaya A. Mmonu, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Nnenaya.Mmonu@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.